CLINICAL TRIAL: NCT03880253
Title: A Placebo-Controlled, Double-Blind, Multiple Ascending Dose Study to Evaluate the Safety and Pharmacokinetic Profile of CTP-692 in Healthy Volunteers
Brief Title: Multiple Ascending Dose Study of CTP-692 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: CP692.1003
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CTP-692 Low Dose or Matching Placebo (Experimental): Once daily dosing
  Interventions: Drug: CTP-692
- CTP-692 Mid Dose or Matching Placebo (Experimental): Once daily dosing
  Interventions: Drug: CTP-692
- CTP-692 High Dose or Matching Placebo (Experimental): Once daily dosing
  Interventions: Drug: CTP-692

INTERVENTIONS:
Drug: CTP-692 — Placebo or CTP-692

SUMMARY:
This study will assess in healthy male and female subjects the safety and pharmacokinetic (PK) profiles of 3 dose levels of CTP-692 following 7 days of dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females between 18 and 55 years of age, inclusive
* Body weight ≥ 55 kg and body mass index within the range of 18 to 32 kg/m2, inclusive

Exclusion Criteria:

* Screening laboratory measurements outside the normal range associated with potential risk for the treatment under investigation at screening and/or prior to the first dose of study drug
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen or hepatitis C virus antibody
* History of clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal (GI) conditions
* Positive drug or alcohol test at screening or prior to the first dose of study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety | Assessments done Day 1 - 9
Measurement of CTP-692 exposure in plasma | Assessments done Day 1 - 9

CONTACTS AND LOCATIONS:
Locations (1):
- Collaborative Neuroscience Network, LLC, Long Beach, California, United States